CLINICAL TRIAL: NCT06336733
Title: Randomized Controlled Trial in Patients on Long-term Colchicine With Colchicine-resistant Familial Mediterranean Fever (FMF) to Evaluate the Efficacy of On-demand Anakinra Treatment for Painful Attacks in Patients Who Refuse Continuous Daily Therapy
Acronym: KIN-ATTACK-FMF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220828
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: FMF
Keywords: Anakinra; Familial Mediterranean fever; Colchicine resistance; Randomized prospective study
MeSH Terms: conditions — Familial Mediterranean Fever | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ANAKINRA on Demand (Experimental): On demand Anakinra 100 mg/j from the prodromal phase of the attack until 24 hours of remission (during 7 days maximum) + colchicine + on demand analgesics
  Interventions: Drug: ANAKINRA
- Standard of Care (No Intervention): Usual analgesics + colchicine

INTERVENTIONS:
Drug: ANAKINRA — On demand Anakinra 100 mg/j from the prodromal phase of the attack until 24 hours of remission (during 7 days maximum) + colchicine + on demand analgesics
  Arms: ANAKINRA on Demand

SUMMARY:
To evaluate the efficacy on clinical symptoms in case of FMF attack among FMF patients resistant to Colchicine of

* on demand anakinra treatment (100 mg/d from the prodromal phase of the attack until 24 hours of remission (during 7 days maximum) associated with daily colchicine.
* compared to analgesic associated with daily colchicine in patients refusing continuous anti-IL-1 treatment.

DETAILED DESCRIPTION:
KIN-ATTACK-FMF will be the first randomized prospective study comparing the efficacy of on-demand anakinra versus standard of care treatment in patients with colchicine resistant symptoms of FMF who refuse continuous daily therapy.

Familial Mediterranean fever (FMF) is the most common monogenic autoinflammatory disease (100,000 people worldwide and 7500 in France). It causes monthly recurrent febrile abdominal pain with a biological inflammatory syndrome.

To prevent FMF attacks and development of inflammatory amyloidosis (IA) daily oral colchicine is the first line recommended treatment. 10 to 15% of patients are resistant to colchicine: persistence of 1attack/month over a period of 3 months (in spite of taking the maximum tolerated dose of colchicine daily). Subcutaneous anti-interleukin 1 biotherapies were recently allowed in France combined to daily oral colchicine for colchicine resistant FMF: anakinra (short-acting anti-IL1 drug, daily) or canakinumab (long acting monoclonal anti IL1 antibody, every 2 months). These treatments cost respectively 30 and 12,000 euros/injection.

If abdominal attacks are controlled by colchicine, patients still suffer from lower limb pains, particularly erysipelas like erythema and exertional myalgias, which are very disabling and require use of analgesics or anti-inflammatory. However, in the referral center, 20% of colchicine resistant FMF patients don't receive chronic anti IL1 treatment, despite an indication. Main reasons are: 1-they do not want to inject themselves every day (for anakinra); 2-women of childbearing age are afraid about the impact of biotherapies on their fetus; 3-some do not want to ask for 100% coverage because of the biotherapy cost; 4- the authorization for anti IL1 in FMF is very recent and they want more certainty about its effectiveness.

The hypothesis of the study is that on-demand use of Anakinra from onset of attack until 24 hours of remission (during 7 days maximum) associated with chronic daily colchicine as background treatment in case of attack could stop it, thus reducing its length and pain compared to standard of care treatment which includes only classical antalgics with colchicine in patients refusing chronic daily anti IL1 treatment.

In the experimental arm, patients receive on demand anakinra treatment (100 mg/d from the prodromal phase of the attack until 24 hours of remission (during 7 days maximum) associated with daily colchicine. In the control arm, patients receive analgesics associated with daily colchicine.

50 participants should be included in the study during a period of 24 months with a 6 months participation period (treatment + follow up)

It's a Multicenter national study including 11 centers.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 6 years old with no upper limit
* Proven FMF according to Livneh international criteria and 2 non ambiguous MEFV mutations.
* Colchicine resistance defined as persistent FMF attack despite the maximum daily posology of colchicine (average one or more attacks per month over a 3-months period)

FMF Attack is defined by:

* Arthritis or
* Chest pain or
* Abdominal pain or
* Myalgia or
* Erysipelas-like skin lesion Duration of episodes 1-4 days.
* Patient refusing daily anakinra injections-
* Patients covered at 100% by the health insurance (ALD)
* Patient who do not have biological inflammation between attacks
* Written informed consent of the patients and or his legal representatives

Exclusion Criteria:

* Evidence of active tuberculosis
* Infection requiring treatment with intravenous antibiotics within 2 weeks prior to inclusion
* History of recurrent infection (Need more than 4 courses of antibiotic treatment per year (in children) or more >2 times per year (in adults), experience pneumonia twice over any time or >3 bacterial sinusitis in 1 year)
* Contraindication to anakinra (Hypersensitivity to the active substance or to any of the excipients (Citric acid, anhydrous Sodium chloride, Disodium edetate dehydrate, Polysorbate 80, Sodium hydroxide, Water for injections ) or to E. coli derived proteins
* Patients with neutropenia (ANC <1.5 x 10^9/l)
* Inability to provide informed consent
* Ongoing chronic treatment with anti IL1 biotherapy since at least 3 months
* Pregnant women
* Women in labor and nursing mothers
* Patients in emergency situations and people hospitalized without consent
* No health care insurance
* Contraindication to colchicine
* Patient participating in another interventional clinical trial
* Patient deprived of liberty
* Patient under guardianship or curatorship
* Patient under court protection

Randomization criteria :

* Absence of active or latent tuberculosis (no tuberculosis sign on chest X-ray and a negative quantiferon)
* Negative pregnancy test

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-12-04 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
Mean number of FMF-attacks per month at 6 months of treatment. | At Months 0 (baseline), Month 1, Month 3 and Month 6
  * FMF attacks is defined by a painful (consensual definition) manifestation during 12 to 72 hours, in either :
    * abdomen (with features consistent with a diagnosis of peritonitis),
    * chest (with features consistent with a diagnosis of pleuritis),
    * joints (with features consistent with a diagnosis of lower extremity large joint monoarthritis),
    * skin (with features consistent with a diagnosis of erysipeloid rash)
  * The painful manifestation can be (or not) accompanied by fever of ≥ 38°C Patients will be asked to note the number of days of pain of each inflammatory attack on a diary.

SECONDARY OUTCOMES:
Cumulative days of FMF attack treatment from randomization to 6 months | At Months 0 (baseline), Month 1, Month 3 and Month 6
  The number of days of injections (for anakinra arm) or number of days of consumption of analgesics (for control group) will be collected via a notebook . Safety
AIDAI (Auto-inflammatory Diseases activity index) score | At Months 0 (baseline), Month 1, Month 3 and Month 6
  Patients will complete the AIDAI (Auto-inflammatory Diseases activity index) score monthly.
Number of painful days and severity of FMF attacks occurring between randomization and M6 | At Months 0 (baseline), Month 1, Month 3 and Month 6
  Number of painful days will be measured by VAS (Visual Analogue Scale) and collected via a notebook).
Quality of life score measured by EuroQOL questionnaire (EQ-5D5L) | At Months 0 (baseline), Month 1, Month 3 and Month 6
  The EQ5D5L will be completed at each visit
Number of local cutaneous reactions at 6 months (erythema and oedema involving the injection sites) in the anakinra arm | At Months 0 (baseline), Month 1, Month 3 and Month 6
  Number of local cutaneous reaction will be collected via a notebook
Proportion of Adverse events | At Months 0 (baseline), Month 1, Month 3 and Month 6
  Adverse events will be collected via a notebook

CONTACTS AND LOCATIONS:
Overall Officials: Léa Léa Léa SAVEY, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Médecine interne Hopital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables,figures, and appendices) could be shared.
  Data would be available Beginning 9 months and ending 36 months following article publication with Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose for individual participant data meta-analysis.
  Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.